CLINICAL TRIAL: NCT06892938
Title: Finger Worn Detection Via Electrocardiographic Ring of Atrial Fibrillation and ECG Waveform Analysis (FINDER-AF)
Brief Title: Detection and Classification of Cardiac Rhythm and Atrial Fibrillation Using a Finger-worn Ring
Acronym: FINDER-AF
Status: Active, not recruiting | Type: Observational
Sponsor: Everbeat (Industry)
Responsible Party: Sponsor
Other Study IDs: EVB002
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF); Arrhythmias Cardiac; Tachycardia; Palpitations; Bradycardia
Keywords: Atrial Fibrillation; Wearable Monitor; Electrocardiogram; Ring
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Tachycardia; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Atrial Fibrillation history: Atrial fibrillation history or active atrial fibrillation
  Interventions: Diagnostic Test: Atrial Fibrillation Identification
- Normal heart rhythm: Patients with no history of prior or active heart arrhythmia
  Interventions: Diagnostic Test: Atrial Fibrillation Identification

INTERVENTIONS:
Diagnostic Test: Atrial Fibrillation Identification — Identification of atrial fibrillation by device.

SUMMARY:
Everbeat is a finger-worn ring that has a built-in electrocardiogram (ECG). In this study the investigators ensure that the ECG as read by the everbeat correctly classifies heart rhythms and detects atrial fibrillation. Investigators will also correlate the everbeat ECG waveform with a clinical-grade FDA approved electrocardiogram to ensure it may be reliably interpreted by clinicians or other algorithms.

DETAILED DESCRIPTION:
In this study the participant will obtain a simultaneous electrocardiogram from both the everbeat ring system and a clinical-grade diagnostic ECG machine for correlation and analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Presence of pacemaker or defibrillator
* Inability to wear a ring in size range available

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with or without cardiac arrhythmic history who are 18 years or older and do not have an implanted cardiac device.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Rhythm classification | Baseline
  Automated rhythm characterization by the ring device as normal sinus rhythm, atrial fibrillation or other.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Civello, MD, Principal Investigator — Our Lady of Lake Hospital
Locations (3):
- United States (3):
  - XIMED, La Jolla, California
  - Our Lady of Lake Hospital, Baton Rouge, Louisiana
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Single study